CLINICAL TRIAL: NCT02633215
Title: Enhancing Cortical Plasticity With Nerve Stimulation in Stroke Patients With Severe Motor Deficit
Brief Title: Enhancing Plasticity in Stroke Patients With Severe Motor Deficit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumy Sawaki (Other)
Responsible Party: Sponsor-Investigator, Lumy Sawaki, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0530242N
Record Dates: First submitted 2015-12-11; First posted 2015-12-17 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: motor recovery; neuroplasticity; chronic; human; sensory
MeSH Terms: conditions — Stroke; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active stimulation with motor training (Experimental): 2 hours of active peripheral nerve stimulation (intervention) paired with 4 hours of intensive task-oriented upper extremity training. Peripheral nerve stimulation of Erb's point, radial and median nerves paired with task-oriented therapy. Peripheral nerve stimulation will be delivered using a S88 Dual Output Stimulator by Grass Technologies.
  Interventions: Device: S88 Dual Output Stimulator by Grass Technologies
- Sham stimulation with motor training (Active Comparator): 2 hours of sham peripheral nerve stimulation (intervention) paired with 4 hours of intensive task-oriented upper extremity training. Peripheral nerve stimulation of Erb's point, radial and median nerves paired with task-oriented therapy. Peripheral nerve stimulation will be delivered using a S88 Dual Output Stimulator by Grass Technologies.
  Interventions: Device: S88 Dual Output Stimulator by Grass Technologies

INTERVENTIONS:
Device: S88 Dual Output Stimulator by Grass Technologies — Peripheral nerve stimulation of Erb's point, radial and median nerves paired with task-oriented therapy

SUMMARY:
This study will evaluate the effectiveness of sustained peripheral nerve stimulation coupled with functional motor training, to improve hand motor function in poorly recovered stroke patients. The central hypothesis is that stroke patients with severe motor deficit receiving hand nerve stimulation and intensive task-oriented therapy will have improved motor function compared to patients receiving sham nerve stimulation and task-oriented therapy.

DETAILED DESCRIPTION:
Stroke is one of the most devastating and prevalent diseases, but efforts to limit the amount of tissue damaged in the acute phase have been disappointing, highlighting the need for effective therapeutic interventions after neurologic damage has occurred. Data from animal and human models have suggested that sensory input plays an important role in motor output, possibly by influencing cortical plasticity. However, in spite of the advances to date, little is known about the extent to which sensory input in the form of peripheral nerve stimulation can be successfully combined to physical training especially in poorly recovered stroke patients. This study will evaluate the effectiveness of sustained peripheral nerve stimulation coupled with functional motor training, to improve hand motor function in stroke patients with severe motor deficit. The central hypothesis is that stroke patients with severe motor deficit receiving hand nerve stimulation and intensive task-oriented therapy will have improved motor function compared to patients receiving sham nerve stimulation and task-oriented therapy, and the degree of this behaviorally-measured effect will correlate with the neurophysiological effect measured by transcranial magnetic stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke patients
* Single stroke
* Chronic (more than 12 months after from stroke)
* At least 21 years old, but there is no upper age range for this project.
* Participants NOT able to extend the affected metacarpophalangeal joints at least 10° and the wrist 20°.

Exclusion Criteria:

* History of carpal tunnel syndrome and conditions that commonly cause peripheral neuropathy, including diabetes, uremia, or associated nutritional deficiencies
* History of head injury with loss of consciousness, severe alcohol or drug abuse, psychiatric illness
* Within 3 months of recruitment, use of drugs known to exert detrimental effects on motor recovery
* Cognitive deficit severe enough to preclude informed consent
* Positive pregnancy test or being of childbearing age and not using appropriate contraception
* Participants with history of untreated depression.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carrico C, Chelette KC 2nd, Westgate PM, Powell E, Nichols L, Fleischer A, Sawaki L. Nerve Stimulation Enhances Task-Oriented Training in Chronic, Severe Motor Deficit After Stroke: A Randomized Trial. Stroke. 2016 Jul;47(7):1879-84. doi: 10.1161/STROKEAHA.116.012671. Epub 2016 May 17. PMID 27188405

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Stimulation With Motor Training | Sham Stimulation With Motor Training
Started | 18 | 18
Completed | 16 | 15
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Stimulation With Motor Training | Sham Stimulation With Motor Training | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (12.1) | 65.4 (10.8) | 62.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Fugl Meyer Assessment Motor Score
Description: Score after intervention minus baseline score, score at 1-month follow-up minus baseline score. The possible scores range from 0 to 66, with 66 indicating the best performance.
Time Frame: baseline, post-intervention, 1-month follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active Stimulation With Motor Training | Sham Stimulation With Motor Training
Number analyzed (Participants) | 18 | 18
units on a scale
  Post-intervention minus baseline | 7.4 (1.0) | 3.4 (1.0)
  1-month follow-up minus baseline | 7.2 (1.3) | 2.8 (1.4)

2. Secondary Outcome: Change in Action Arm Research Test (ARAT)
Description: Score at post-intervention minus baseline, score at 1-month follow-up minus baseline. The possible scores range from 0 to 57, with higher scores indicating better performance.
Time Frame: baseline, post-intervention, 1-month follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active Stimulation With Motor Training | Sham Stimulation With Motor Training
Number analyzed (Participants) | 18 | 18
units on a scale
  Post-intervention minus baseline | 6.4 (1.1) | 2.3 (1.1)
  1-month follow-up minus baseline | 6.9 (1.3) | 2.4 (1.4)

3. Secondary Outcome: Change in Wolf Motor Function Test (WMFT)
Description: Score at post-intervention minus baseline, score at 1-month follow-up minus baseline. Each task is scored as amount of time taken to complete a task, which may range from just over 0 to 120 seconds. If the subject is unable to complete the task within 120 seconds, a score of 121 seconds is given. The scores from the 15 individual tasks are averaged, then the log is taken, resulting in the overall score. Therefore, the larger the score, the longer required to perform the tasks. Negative changes in score indicate that a subject, on average, was able to complete the tasks faster at post-intervention or at 1-month follow-up than at baseline.
Time Frame: baseline, post-intervention, 1-month follow-up
Measure: Mean (Standard Error); unit: log(seconds)
Arm/Group | Active Stimulation With Motor Training | Sham Stimulation With Motor Training
Number analyzed (Participants) | 18 | 17
log(seconds)
  Post-intervention minus baseline | -0.18 (0.03) | -0.06 (0.03)
  1-month follow-up minus baseline | -0.14 (0.03) | -0.07 (0.04)

ADVERSE EVENTS:
Arm/Group | Active Stimulation With Motor Training | Sham Stimulation With Motor Training
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No